CLINICAL TRIAL: NCT00470600
Title: A MULTI-CENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED TRIAL OF IBUPROFEN INJECTION (IVIb) FOR TREATMENT OF PAIN IN POST-OPERATIVE ORTHOPEDIC ADULT PATIENTS
Brief Title: Efficacy and Safety Study of Caldolor (IV Ibuprofen) in Hospitalized Adult Orthopedic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPI-CL-008C
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ibuprofen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal Saline (Placebo Comparator): 250 milliliters normal saline as a placebo comparator was administered every 6 hours for a total of five doses over the first 24 hours. Those patients who received the initial five doses could continue to receive additional doses as needed every 6 hours through the 120-hour treatment period.
  Interventions: Other: Normal Saline
- Intravenous ibuprofen (Experimental): 800 mg of intravenous ibuprofen diluted in 250 milliliters normal saline was administered every 6 hours for a total of five doses over the first 24 hours. Those patients who received the initial five doses could continue to receive additional doses as needed every 6 hours through the 120-hour treatment period.
  Interventions: Drug: Caldolor

INTERVENTIONS:
Drug: Caldolor — 800 milligrams intravenous
  Other Names: Ibuprofen
  Arms: Intravenous ibuprofen
Other: Normal Saline — Placebo comparator
  Other Names: NS
  Arms: Normal Saline

SUMMARY:
The primary objective of this study of Caldolor (IV ibuprofen) administered to post-operative hospitalized adult orthopedic patients every 6 hours for at least 24 hours is to determine the efficacy of Caldolor (IV ibuprofen) compared to placebo for the treatment of post-operative pain by patients self-assessment of pain.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for elective hip or knee replacement, reconstruction or arthroplasty surgery with anticipated need for post-operative intravenous (IV) morphine analgesia with anticipated use of (greater than or equal to (≥) 28 hours.
2. Adequate IV access
3. Anticipated hospital stay ≥ 28 hours

Exclusion Criteria:

1. Be unable to make a reliable self-report of pain intensity to pain relief
2. Less than 18 years of age
3. Greater than 80 years of age
4. Use of analgesics, muscle relaxants, NSAIDS and sedatives less than 12 hours prior to clinicaltrial material(CTM) administration with the following exceptions: paracetamol (acetaminophen) can be administered until 6 hours prior to surgery; tramadol can be administered until midnight the evening prior to surgery; muscle relaxants working at the neuromuscular junction used for intubation and/or anesthesia administration for the surgical procedure prior to CTM administration; and sedatives (i.e., midazolam) used as a co-induction agent for the surgical procedure prior to CTM administration
5. Patients taking warfarin, lithium, combination of angiotension converting enzyme(ACE)-inhibitors and furosemide
6. Patients with anemia (active, clinically significant anemia) and/or a history or evidence of asthma or heart failure
7. History of allergy or hypersensitivity to any component of Caldolor, aspirin (or aspirin related products), NSAIDs, or COX-2 inhibitors
8. Pregnant or nursing
9. History of severe head trauma that required current hospitalization, intracranial surgery or stroke within the previous 30 days, or any history of intracerebral arteriovenous malformation, cerebral aneurysm or CNS mass lesion
10. Weigh less than 30 kilogram
11. Have a history of congenital bleeding diathesis (e.g. hemophilia) or any active clinically significant bleeding, or have underlying platelet dysfunction including (but not limited to) idiopathic thrombocytopenic purpura, disseminated intravascular coagulation, or congenital platelet dysfunction
12. Have gastrointestional (GI) bleeding that required medical intervention within the previous 6 weeks (unless definitive surgery has been performed)
13. Have a platelet count less than 30,000 mm^3 determined within the 28 days prior to surgery
14. Pre-existing dependence on narcotics or known tolerance to opioids
15. Inability to understand the requirements of the study, be willing to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]), and agree to abide by the study restrictions and to return for the required assessments
16. Refusal to provide written authorization for use and disclosure of protected health information
17. Be on dialysis, have oliguria or creatinine greater than 3.0 milligram/deciliter.
18. Inability to achieve hemostasis or inability to close surgical incision, prior to Operating Room discharge
19. Operative procedure includes organ transplant
20. Pre or intra-operative procedure utilized for the prevention of pre- or post-operative pain (i.e. epidural or nerve blocks)
21. Be receiving full dose anticoagulation therapy or Activated Protein C within 6 hours before dosing (Prophylaxis with subcutaneous heparin is acceptable)
22. Have received another investigational drug within the past 30 days
23. Be otherwise unsuitable for the study in the opinion of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2007-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Singla, MD, Principal Investigator — Lotus Clinical Research/Methodist Hospital of Southern CA
Locations (9):
- United States (6):
  - Wilmax Clinical Research Inc., Mobile, Alabama
  - Teton Research, LLC, Little Rock, Arkansas
  - Clinical Management Services, Inc., Arcadia, California
  - Southeastern Center for Clinical Trials, Atlanta, Georgia
  - Research Concepts, Inc, Houston, Texas
  - Research Concepts, Inc., Houston, Texas
- South Africa (3):
  - Johannesburg General Hospital, Johannesburg
  - Krugersdorp Private Hospital, Krugersdorp
  - Eugene Marais Hospital, Pretoria

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 250 mL of normal saline.
- 800mg IV Ibuprofen (Caldolor): 8 mL of IV Ibuprofen (Caldolor) added with 250 mL of normal saline to give 800 mg dose.
Period: Overall Study
Arm/Group | Placebo | 800mg IV Ibuprofen (Caldolor)
Started | 86 | 99
Completed | 86 (Two subjects were randomized to incorrect stratification categories (weight).) | 99 (One subject was randomized to incorrect stratification categories (weight).)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 800mg IV Ibuprofen (Caldolor) | Total
Number analyzed (Participants) | 86 | 99 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (9.9) | 62 (10.3) | 61 (10.2)
Age, Customized [Number; unit: participants]
  <45years | 6 | 3 | 9
  >= 45 years | 80 | 96 | 176
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 65 | 120
  Male | 31 | 34 | 65
Region of Enrollment [Number; unit: participants]
  United States | 61 | 70 | 131
  South Africa | 25 | 29 | 54

OUTCOME MEASURES:

1. Primary Outcome: AUC-VAS With Movement (Post-operative Period, Hour-6-28)
Description: Measurement of the patient's self assessment of pain with movement using the validated visual analog scale (VAS) during the post-operative period (study hour-6 through hour-28). VAS assessments document the patient's self reported level of pain from "No pain" (0 mm) to "Worst possible pain" (100 mm) on a 100 mm line. VAS assessments were performed immediately following surgery [variable since every surgery has a unique length of time even if it is the same procedure] and at hours 6, 8, 12, 16, 20, 24 and 28 (for the primary endpoint).
Time Frame: Study hour-6 through hour-28
Population: Efficacy analyses were performed on the Intent to Treat (ITT) population and the Efficacy Evaluable Population (EEP). All randomized patients who received at least a partial dose of CTM were included in the ITT analyses. All data below represents the ITT analyses.
Measure: Least Squares Mean (Standard Error); unit: AUC-VAS pain v. time (mm*hr)
Arm/Group | Placebo | 800mg IV Ibuprofen (Caldolor)
Number analyzed (Participants) | 84 | 95
AUC-VAS pain v. time (mm*hr) | 1326.1 (82.0) | 1005.0 (81.5)

2. Secondary Outcome: Secondary Endpoint: AUC-VAS at Rest (Post-operative Period, Hours 6-28)
Description: Measurement of the patient's self assessment of pain at rest using a visual analog scale (VAS) during the post-operative period (study hour-6 through hour-28). VAS assessments document the patient's self reported level of pain from "No pain" (0 mm) to "Worst possible pain" (100 mm) on a 100 mm line. VAS assessments were performed immediately following surgery and at hours 6, 8, 12, 16, 20, 24 and 28 (for the primary endpoint).
Time Frame: Study hour-6 through hour-28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: AUC-VAS pain v. time (mm*hr)
Arm/Group | Placebo | 800mg IV Ibuprofen (Caldolor)
Number analyzed (Participants) | 84 | 95
AUC-VAS pain v. time (mm*hr) | 997.0 (83.6) | 728.0 (83.0)

3. Secondary Outcome: Patient Demand of Narcotic Use (Post-operative Period, From Hour 6 to 28).
Description: Patient demand of narcotic used by patients in each treatment group for analgesia, post-surgery.
Time Frame: Study hour-6 to hour-28
Population: Demand of narcotic use was determined by PCA records or by chart if patient requested and not via PCA.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Placebo | 800mg IV Ibuprofen (Caldolor)
Number analyzed (Participants) | 84 | 95
milligrams | 59.5 (29.9) | 41.1 (27.3)

ADVERSE EVENTS:
Arm/Group | Placebo | 800mg IV Ibuprofen (Caldolor)
Serious Adverse Events (participants affected / at risk) | 3/86 | 8/99
Other Adverse Events (participants affected / at risk) | 74/86 | 90/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=86) | 800mg IV Ibuprofen (Caldolor) (N=99)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Post procedural pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Altered mental status (Psychiatric disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=86) | 800mg IV Ibuprofen (Caldolor) (N=99)
Vomiting (Gastrointestinal disorders) | 12 (13) | 27 (28)
Constipation (Gastrointestinal disorders) | 11 (11) | 20 (20)
Dyspepsia (Gastrointestinal disorders) | 4 (5) | 0 (0)
Body temperature increased (Investigations) | 11 (11) | 8 (10)
Urine output decreased (Investigations) | 8 (9) | 5 (5)
Haemaglobin decreased (Investigations) | 0 (0) | 4 (4)
Pyrexia (General disorders) | 15 (16) | 14 (18)
Oedema Peripheral (General disorders) | 2 (2) | 3 (6)
Pruritis (Skin and subcutaneous tissue disorders) | 17 (22) | 10 (13)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 6 (6) | 8 (9)
Hypertension (Vascular disorders) | 3 (3) | 3 (4)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 10 (10) | 10 (10)
Urinary retention (Renal and urinary disorders) | 2 (2) | 9 (10)
Dysuria (Renal and urinary disorders) | 5 (6) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 5 (7) | 3 (4)
Dizziness (Nervous system disorders) | 3 (4) | 4 (4)
Insomnia (Psychiatric disorders) | 2 (2) | 7 (7)
Agitation (Psychiatric disorders) | 1 (1) | 3 (3)
Tachycardia (Cardiac disorders) | 3 (3) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 30 (37) | 44 (47)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No